CLINICAL TRIAL: NCT07039292
Title: A Novel Harm Reduction Approach for Oncology Outpatients Who Smoke and Refuse Traditional Tobacco Treatment
Brief Title: Clinical Alternatives for Reducing Harm Using E-cigarettes
Acronym: CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Alana Rojewski, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00138162; 1R01CA293735-01A1 (NIH)
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Smoking; E-Cig Use; Oncology
MeSH Terms: conditions — Smoking; Vaping; Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Harm Reduction (E-cigarette switching) (Experimental): Participants will be assigned to receive an e-cigarette and try to switch completely from smoking to using the e-cigarette
  Interventions: Behavioral: Harm Reduction (E-cigarette switching)
- Standard of Care (Active Comparator): Participants will be assigned to receive tobacco treatment referrals and the opportunity to re-enroll in the Tobacco Treatment Program
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Harm Reduction (E-cigarette switching) — Participants will be assigned to receive an e-cigarette and try to switch completely from smoking to using the e-cigarette
  Arms: Harm Reduction (E-cigarette switching)
Behavioral: Standard of Care — Participants will be assigned to receive tobacco treatment referrals and the opportunity to re-enroll in the Tobacco Treatment Program
  Arms: Standard of Care

SUMMARY:
For patients in cancer care, quitting smoking is critical, but a significant portion of patients in cancer care refuse all components of tobacco treatment, even when offered free of charge. The proposed clinical trial will assess one harm reduction intervention, switching completely from cigarettes to e-cigarettes, among oncology outpatients who smoke and refuse traditional tobacco treatment. This study is a type 1 hybrid effectiveness-implementation trial among oncology outpatients at an NCI-designated cancer center who smoke and refuse all components of tobacco treatment (N=208).

DETAILED DESCRIPTION:
In the proposed study, we will conduct a type 1 hybrid effectiveness-implementation trial (N=208) to directly compare rates of switching to e-cigarettes to standard care, and advance understanding of key barriers and facilitators of implementation processes. Outpatients at HCC clinics who have opted out of traditional tobacco treatment will be randomly assigned to either 1) an e-cigarette switching approach (Switch), or 2) standard of care (SC; provision of additional tobacco treatment resources). We will compare rates of switching between the two groups, and conduct a mixed methods evaluation of implementation processes for the e-cigarette switching approach. To further evaluate the impact of harm reduction in this population, we will also collect exploratory data on the impact of switching to e-cigarettes on the biological effects of cancer risk (i.e., inflammation and DNA damage) and subjective effects of product use on health-related quality of life.

Potential subjects will be recruited and screened for inclusion and exclusion criteria from MUSC's telehealth TTP. Once we have determined that someone meets our eligibility criteria, we will invite them to begin the consent process. Participants who consent to participation and are randomized will complete baseline assessments, a baseline breath CO, and a blood draw for baseline biomarker assessment. Participants in the Switch group will be provided with a 13-week supply of e-cigarettes and choose a switch date.

Participants will be asked to complete Assessments remotely via REDCap survey on the Target Switch Day (Week 0 Assessment), and every 2 weeks through the end of product provision (Week 12). An additional assessment will be completed at the Week 24 follow-up. Participants will complete a blood draw at Baseline, Week 12, and Week 24. Participants will complete a remote submission of breath carbon monoxide at baseline, Week 0 (Switch Date), Week 6, Week 12, and Week 24.

We will conduct semi-structured interviews with ~20-25 participants from Switch after they complete the Week 24 follow-up to gain in-depth understanding of intervention experiences. We will also interview the primary providers from MUSC TTP who conducted the telehealth counseling component as well as other key clinic stakeholders. The providers will be interviewed on intervention acceptability including their perceptions of e-cigarettes as harm reduction tools, reach, fit within the clinic environment, resources to support and sustain the intervention in practice, and implementation barriers and facilitators.

ELIGIBILITY:
Inclusion Criteria:

* age 21+,
* identified as smoking in their medical record and self-report of current smoking within the past 30 days
* refused traditional treatment options through the opt-out HCC Tobacco Treatment Program
* English speaking;

Exclusion Criteria:

* currently taking part in any TTP or using cessation medication (i.e., taking NRT or other cessation medications, enrolled in the Quitline, or in another study),
* use of e-cigarettes in the past 30 days,
* currently imprisoned,
* pregnant women.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Complete switching | 6 months
  The percentage of participants who are abstinent from combustible cigarettes at the 6-month follow up

SECONDARY OUTCOMES:
Implementation | 12 weeks
  Percentage of people who smoke who engage in the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alana Rojewski, Principal Investigator — Medical University of South Carolina; Tracy Smith, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States